CLINICAL TRIAL: NCT03642522
Title: Investigating Predictors of Treatment Response in Treatment-Resistant Depression (TRD) With Interleaved TMS/fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Victoria (Other)
Responsible Party: Principal Investigator, Fidel Vila-Rodriguez, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H14-02819
Record Dates: First submitted 2018-08-09; First posted 2018-08-22 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Major Depressive Disorder; Depression
Keywords: repetitive transcranial magnetic stimulation; rTMS; neurostimulation; biomarker; treatment-resistant
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 Hz rTMS (Experimental): 30 minutes of 1 Hz rTMS to the right dorsolateral prefrontal cortex (R_DLPFC)
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — rTMS is a Health-Canada- and FDA-approved treatment for treatment-resistant depression (TRD), using focused magnetic field pulses to stimulate brain regions involved in emotion regulation, safely and non-invasively. rTMS can be applied at varying discharge frequencies which have differential effects on cortical excitability. At a low frequency (≤ 1Hz), rTMS reduces cortical excitability, while at frequencies greater than 1 Hz, rTMS facilitates cortical excitability3. In MDD, either high- frequency rTMS (HF-rTMS) applied over the left dorsolateral prefrontal cortex (DLPFC) or low- frequency rTMS (LF-rTMS) applied over the right DLPFC have similar efficacy. This study utilizes low frequency rTMS to the right DLPFC.
  Other Names: rTMS

SUMMARY:
The purpose of this trial is identify biomarkers of response to repetitive transcranial magnetic stimulation (rTMS) in individuals with first episode or treatment resistant depression. These biomarkers include simultaneous TMS-fMRI (functional magnetic resonance imaging), a blood smear, cognitive and behavioural assessments, questionnaires, and neurophysiology.

DETAILED DESCRIPTION:
This study is enrolling 60 individuals with treatment-resistant depression.

All patients will receive four weeks of 1-Hz rTMS to the right dorsolateral prefrontal cortex (R_DLPFC). In addition, all patients will undergo baseline and post-treatment measures, including rTMS while they are in the MRI scanner, neurophysiology (Electroencephalography (EEG)/Near-Infrared Spectroscopy (NIRS)), cognitive testing, behavioural assessments and a blood smear. There will also be a 1-week, 4-week, and 12-week follow-up following completion of the treatment course.

ELIGIBILITY:
TRD Patient Inclusion Criteria:

Patients will be included if they:

1. are outpatients
2. are voluntary and competent to consent to treatment
3. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of MDD, single or recurrent
4. are between the ages of 18 and 80 years
5. have failed to achieve a clinical response to at least one adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of score ≥ 3 in the current episode OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF 1 or 2)
6. have a score ≥ 22 on the IDS item
7. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to initiation of rTMS
8. able to adhere to the treatment schedule
9. pass the TMS adult safety screening (TASS) questionnaire

First Episode Depression Inclusion Criteria:

Patients will be included if they:

1. are outpatients
2. are voluntary and competent to consent to treatment
3. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of MDD, single or recurrent
4. are between the ages of 18 and 80 years
5. have never received and adequate antidepressant trial and are not currently taking any antidepressant.
6. have a score ≥ 12 on the IDS item
7. are on no psychotropic medication for the 4 weeks prior to initiation of rTMS, with the exception of lorazepam up to 2mg or equivalent dose of benzodiazepine or prescribed sleeping aids including (zopiclone up to 15mg/d, zolpidem up to 10mg/d).
8. able to adhere to the treatment schedule
9. pass the TMS adult safety screening (TASS) questionnaire

Patient Exclusion Criteria:

Patients are excluded if they:

1. have a history of substance dependence or abuse within the last 3 months
2. have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
3. have active suicidal intent
4. are pregnant
5. have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
6. have a MINI diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, assessed by a study investigator to be primary and causing greater impairment than MDD
7. have a diagnosis of any personality disorder, and assessed by a study investigator to be primary and causing greater impairment than MDD
8. have failed a course of ECT in the current episode or previous episode
9. have received rTMS for any previous indication due to the potential compromise of expectancy effects
10. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than 5 minutes
11. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
12. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
13. have a clinically significant laboratory abnormality, in the opinion of the one of the principal investigators
14. are currently (or in the last 4 weeks) taking lorazepam greater than 2 mg daily (or equivalent) or any dose of an anticonvulsant, due to the potential to limit rTMS efficacy
15. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).
16. have failed more than 5 adequate trials of medication in the current episode.
17. Exclusion criteria for MRI: Those with a history of cranial, thoracic or abdominal surgery, with pacemakers, artificial joins or other metallic implants will be excluded from the MRI scan. Subjects that have agreed to participate in the MRI portion of the study will be pre- screened for any potential metal fragments in the body (particularly in the orbits) if they have had any history of doing metal work or have been involved in use/deployment of ammunitions/explosives, welding, piping etc.). In these cases a CT scan will be performed prior to the MRI scan

    ----------

Healthy Control Inclusion Criteria

Participants will be included if they:

1. are voluntary and competent to consent to the study
2. are between the ages of 18 and 80
3. are fluent in English, sufficient to complete interviews and cognitive testing
4. have no history of Axis I or Axis II disorders, as determined by the MINI
5. pass the TMS adult safety screening (TASS) questionnaire

Healthy Control Exclusion Criteria:

Participants will be excluded if they:

1. have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
2. have a MINI diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), dysthymia or any personality disorder
3. have history of bipolar disorder or psychosis in first degree relative (parents, siblings, offspring)
4. are unable to provide family history of biological family (i.e., adopted persons are not eligible)
5. have a history of substance dependence within the last 3 months
6. have a concomitant major unstable medical illness
7. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
8. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).
9. have a personal or family history of seizures
10. Exclusion criteria for MRI: Those with a history of cranial, thoracic or abdominal surgery, with pacemakers, artificial joins or other metallic implants will be excluded from the MRI scan. Those who are pregnant will also be excluded from the MRI scan. Subjects that have agreed to participate in the MRI portion of the study will be pre-screened for any potential metal fragments in the body (particularly in the orbits) if they have had any history of doing metal work or have been involved in use/deployment of ammunitions/explosives, welding, piping etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology (IDS-30) | 4 weeks
  The inventory of depressive symptomatology is a clinician-rated depression scale. Outcome will be total score. Minimum score is 0 and maximum score is 84. Higher scores indicate worse severity.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology (QIDS-SR) | 4 weeks
  The quick inventory of depressive symptomatology is self-rated depression scale. Outcome will be total score. Minimum score is 0 and maximum score is 27. Higher scores indicate worse severity.

OTHER OUTCOMES:
Quick Inventory of Depressive Symptomatology (QIDS-SR) | 16 weeks
  The quick inventory of depressive symptomatology is self-rated depression scale. Outcome will be total score. Minimum score is 0 and maximum score is 27. Higher scores indicate worse severity.
Inventory of Depressive Symptomatology (IDS-30) | 16 weeks
  The quick inventory of depressive symptomatology is self-rated depression scale. Outcome will be total score. Minimum score is 0 and maximum score is 27. Higher scores indicate worse severity.
The Montgomery-Åsberg Depression Rating Scale (MADRS) | 4 weeks
  The Montgomery-Åsberg Depression Rating Scale is a clinician-rated depression scale. Outcome will be total score. Minimum score is 0 and maximum score is 60. Higher scores indicate worse severity.
The Montgomery-Åsberg Depression Rating Scale (MADRS) | 16 weeks
  The Montgomery-Åsberg Depression Rating Scale is a clinician-rated depression scale. Outcome will be total score. Minimum score is 0 and maximum score is 60. Higher scores indicate worse severity.

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Vila-Rodriguez, MD, Principal Investigator — University of British Columbia
Locations (1):
- Non-Invasive Neurostimulation Therapies lab, University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ge R, Humaira A, Gregory E, Alamian G, MacMillan EL, Barlow L, Todd R, Nestor S, Frangou S, Vila-Rodriguez F. Predictive Value of Acute Neuroplastic Response to rTMS in Treatment Outcome in Depression: A Concurrent TMS-fMRI Trial. Am J Psychiatry. 2022 Jul;179(7):500-508. doi: 10.1176/appi.ajp.21050541. Epub 2022 May 18. PMID 35582784